CLINICAL TRIAL: NCT02110576
Title: Procedure For The Reference Range Study For Absolute MA
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100343
Record Dates: First submitted 2014-03-28; First posted 2014-04-10 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Transmission, Blood, Recipient/Donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Controls: Healthy controls in general good health, without chronic disease/illness, including but not limited to: cancer, diabetes mellitus, renal disease, cardiac disease, hypertension, lung disease, liver disease, complications of morbid obesity, autoimmune/inflammatory disease, or any condition of sufficient severity that it requires daily medication to manage

SUMMARY:
CLSI guidelines shall be followed to gather data from a minimum of one hundred and twenty normal donors to create reference intervals for various Haemonetics reagents. Venous blood from a minimum of 146 reference subjects shall be tested. Blood from 160 donors will be drawn at the study site to account for aberrant or outlying data excluded for technical or other reasons.

DETAILED DESCRIPTION:
As part of an examination of how LY30 is calculated, the investigators would like to explore the differences between Maximum Amplitude (MA) and LY30 calculated in the traditional small deviation method and by an absolute MA method.

The maximum amplitude (MA) for a sample is determined in real-time using one of two MA-identifying algorithms: Small Deviation MA (the default algorithm) or Absolute MA. Both algorithms are available in commercially available software. Both algorithms find an MA for a sample; however, the difference between the two algorithms is the "acceptance criteria" which each use for identifying the MA. As compared to Small Deviation MA, the Absolute MA has a larger and more stringent rules set.

A study will be run to establish reference intervals following the guidelines set out in CLSI document C28-A3c. This guideline calls for a reference interval to be constructed from at least 120 donors. To meet the guidance outlined in the CLSI guideline, we will collect a minimum of 146 donors.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over the age of 18 years.
* Self-identified as being in general good health, without chronic disease/illness, including but not limited to: cancer, diabetes mellitus, renal disease, cardiac disease, hypertension, lung disease, liver disease, complications of morbid obesity, autoimmune/inflammatory disease, or any condition of sufficient severity that it requires daily medication to manage

Exclusion Criteria:

* Age < 18 years.
* Infusion of blood products prior to the collection of blood samples.
* Known or subsequently discovered inherited defects of coagulation function (e.g. hemophilia or Von Willebrand's disease).
* Those females known to be pregnant
* Anticoagulant, antiplatelet, hormone or hormonal contraceptive therapy including aspirin use within the past month or NSAID use within the past week
* Surgery or traumatic injury within the previous 6 weeks
* Bruising, wounds or scarring in the area of venipuncture on the upper extremities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
TEG Reference Ranges | Up to four months
  Reference ranges will be completed on 50 parameters sample type combinations for which 160 donors will be enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E. Moore, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States